CLINICAL TRIAL: NCT05404555
Title: Prognostic Value of Right Ventricular Myocardial Strain in Patients With Acute Myocardial Infarction With Different Infarction-related Vessels
Brief Title: Prognostic Value of Right Ventricular Myocardial Strain in Patients With Acute Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022093
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-03

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acute myocardia infarction patients with right coronary artery occlusion
  Interventions: Other: two-dimensional speckle tracking echocardiography
- acute myocardia infarction patients with non-right coronary artery occlusion
  Interventions: Other: two-dimensional speckle tracking echocardiography

INTERVENTIONS:
Other: two-dimensional speckle tracking echocardiography — Two-dimensional speckle tracking echocardiography is used to assess cardiac function in all enrolled patients

SUMMARY:
For a long time, the right ventricle has been the "forgotten chamber", but with the deepening of people's understanding of the disease, right ventricular dysfunction has become an important factor to evaluate the disease progression and late prognosis of patients with AMI. Right ventricular myocardial strain derived from two-dimensional speckle tracking echocardiography is a new method for early evaluation of regional and global right ventricular systolic function, and its repeatability is much higher than that of LVEF. Acute inferior myocardial infarction is often caused by occlusion of the proximal middle segment of the right coronary artery. Many studies have confirmed that RVMS is an independent predictor of poor prognosis in patients with AIMI. However, 60% of the right ventricular systolic function is contributed by the left ventricle and interventricular septum, and the left anterior descending branch and the left circumflex branch are the main sources of blood supply to the left ventricle and interventricular septum, so in theory, non-RCA occlusion can also lead to varying degrees of right ventricular dysfunction. However, there are few studies on the role of RVMS in predicting the prognosis of AMI patients caused by non-RCA occlusion. Therefore, the purpose of this study is to prospectively study the value of dynamic changes of RVMS in predicting the prognosis of patients with acute myocardial infarction with different infarct-related vessels, in order to provide more clinical reference information for the diagnosis and treatment of AMI.

DETAILED DESCRIPTION:
In this study, 200 patients with acute myocardial infarction treated in Peking University Third Hospital from March 2022 to March 2024 were enrolled in this study. the parameters of myocardial enzymes, blood lipids and echocardiography were collected at the acute stage, 2 weeks and 6 months after discharge, and were followed up for two year. The echocardiographic parameters and MACE of patients with acute myocardial infarction with different infarction related vessels were compared. This shows the significance of right ventricular myocardial strain in predicting the prognosis of patients with acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females were between 35 and 85 years old;
2. coronary artery disease underwent emergency PCI for NSTEMI or primary PCI for STEMI;
3. coronary artery type was right coronary dominance;
4. regular follow-up for 2 year.

Exclusion Criteria:

1. Patients who cannot complete 2D speckle tracking imaging;
2. patients with severe valvular disease, cardiomyopathy, or congenital heart disease; severe liver and kidney insufficiency or chronic respiratory disease;
3. previous PCI or CABG;
4. coronary artery type: Left crown dominance.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with acute myocardial infarction undergoing primary percutaneous coronary intervention are included.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 2 years
  Nonfatal stroke, nonfatal myocardial infarction, target vessel requiring revascularization, death

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No